CLINICAL TRIAL: NCT04079413
Title: An Open-label, Randomized, Multi-center, Parallel-group Clinical Trial Comparing the Efficacy and Safety of GP40071 (OOO "GEROPHARM", Russia) Compared to NovoRapid® Penfill® (Novo Nordisk A/S, Denmark) in Type 1 Diabetes Mellitus Patients
Brief Title: Efficacy and Safety of GP40071 Compared to NovoRapid® Penfill® in Type 1 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP40071-P4-31
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2019-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
Keywords: Insulin; Insulin aspart; Aspart
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Aspart

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP40071 (Experimental): Subcutaneous (SC), before meals intake, up to Week 26
  Interventions: Drug: GP40071
- NovoRapid® Penfill® (Active Comparator): Subcutaneous (SC), before meals intake, up to Week 26
  Interventions: Drug: NovoRapid® Penfill®

INTERVENTIONS:
Drug: GP40071 — GP40071, 100 per milliliters (U/mL) (dose range of 1 unit to 80 units) self-administered by SC injection, immediately (within 5-10 minutes) before meal intake.
  Other Names: Insulin aspart
  Arms: GP40071
Drug: NovoRapid® Penfill® — NovoRapid® Penfill®, 100 per milliliters (U/mL) (dose range of 1 unit to 80 units) self-administered by SC injection, immediately (within 5-10 minutes) before meal intake.
  Other Names: Insulin aspart
  Arms: NovoRapid® Penfill®

SUMMARY:
This trial is a multi-center, open-label, randomized, parallel group trial in adult patients with T1DM comparing the efficacy and safety of GP40071 (insulin aspart, GEROPHARM) with that of NovoRapid®.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent
* Diabetes mellitus type 1 for at least 12 months prior to screening
* History of basis-bolus (multiple dose injection (MDI)) therapy in stable doses at least 30 days
* Glycated hemoglobin (HbA1c) level of 7.1 to 12.0 % at screening (both values inclusive)
* Body mass index (BMI) of 18.5 to 35 kg/m2 at screening (both values inclusive)
* Subject is able and willing to comply with the requirements of the study protocol

Exclusion Criteria:

* Contraindication to the use of insulin aspart
* Insulin resistance over 1.5 U/kg insulin pro day
* Change INN of insulin for 6 months prior to randomisation
* History of treatment any biosimilar insulin for 6 months prior to randomisation (excl. GEROPHARM's insulins)
* History of treatment any experimental drugs or medical devices for 3 months prior to randomisation
* History of treatment insulin pump for 180 days prior to signed written consent or indication for use insulin pump
* Presence of severe diabetes complications
* History of severe hypoglycemia for 6 months prior to screening
* History of 15 or more episodes mild hypoglycemia for 1 month prior to screening
* History or presence of uncontrolled diabetes mellitus for 6 months prior to screening
* History of administration of glucocorticoids (14 days or more) for 1 year prior to screening
* Administration of any immunosuppressive drugs (Cyclosporine, Methotrexate, Rituximab, etc.)
* History of vaccination for 6 months prior to randomisation
* History of autoimmune disease, except vitiligo and controlled autoimmune polyglandular syndrome (APS) types 1-3, except adrenal insufficiency
* History of unstable angina, myocardial infarction, severe arrhythmia, heart failure III or IV NYHA for 1 year prior to screening
* History of stroke or TIA for 6 months prior to screening
* History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analogue preparations used in the trial, OR history of significant allergic drug reactions
* Pregnant and breast-feeding women
* Acute inflammation disease for 3 weeks prior to screening
* Deviation of the laboratory results conducted during the screening:

Hemoglobin value < 9,0 g/dl; Hematocrit value < 30 %; ALT and AST value > 2 folds as high as maximal normal value; Serum bilirubin value > 1.5 folds as high as maximal normal value

* History of hematological disorders that can affect the reliability of HbA1c estimation (hemoglobinopathies, hemolytic anemia, etc.)
* Serious blood loss for 3 months prior to screening (blood donation, surgery procedure, etc.)
* Incomplete recovery after surgery procedure
* History of drug, alcohol abuse for 3 years prior to screening
* Serological evidence of human immunodeficiency virus (HIV), hepatitis B (HbSAg), hepatitis C (HCVAb) or syphilis (Treponema pallidum) antibodies at screening
* History of oncological disease during 5 years prior to screening
* History of transplantation, except 3 months after corneal transplant
* History or presence of a medical condition or disease that in the investigator's opinion would embarrass glycemic control and completion of the study
* Inability follow to protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 26 weeks
  Change from baseline in titer of antibodies to human insulin

SECONDARY OUTCOMES:
Glycated hemoglobin | 26 weeks
  Change in HbA1c from baseline
Adverse Events frequency and degree | 26 weeks
  Hypoglycemic episodes (glucose level < 3.9 mmol/l) frequency; Occurrence of local reactions at injection sites; Occurrence allergic reactions
Fasting Plasma Glucose Level | 26 weeks
  Change in fasting plasma glucose level from baseline
Seven-Point Glucose Testing | 26 weeks
  Change in seven-point glucose testing results from baseline
Total Insulin Dose | 26 weeks
  Change in total insulin dose per body weight (U/kg) from baseline
Body Mass Index | 26 weeks
  Change in BMI from baseline
Treatment Satisfaction | 26 weeks
  Change in treatment satisfaction from baseline. The total score DTSQ (The Diabetes Treatment Satisfaction Questionnaire) (range 0-36). Questions 1, 4, 5, 6, 7 and 8 assesses treatment satisfaction (summed these 6 questions). Questions 2 and 3 assess the burden from hyper- and hypoglycemia.
Achievement of Glycated Hemoglobin Goals | 26 weeks
  The frequency of achievement glycated hemoglobin goals
Achievement of Glycated Hemoglobin < 7% | 26 weeks
  The frequency of achievement glycated hemoglobin < 7% ( 7% inclusive)

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Kazan Endocrinology Dispensary, Kazan'
  - Krasnoyarsk State Medical University named after Professor V.F. Voino-Yasenetsky, Krasnoyarsk
  - Endocrinology Research Centre (Moscow), Moscow
  - Rostov State Medical University, Rostov-on-Don
  - Polyclinic Сomplex, Saint Petersburg
  - City Diagnostic Center № 1, Saint Petersburg
  - City Polyclinic № 117, Saint Petersburg
  - EosMed, Saint Petersburg
  - Institute of Medical Research, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Pokrovskaya Municipal Hospital, Saint Petersburg
  - Diabetes Center, Samara
  - Clinical City Hospital № 9, Saratov

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Karonova TL, Mayorov AY, Magruk MA, Zyangirova ST, Grigoryeva IV, Khmelnitski OK, Myshkovets A, Parfenova TM, Mosikian AA, Drai RV. Safety and efficacy of GP40071 compared with originator insulin aspart (NovoRapid(R) Penfill(R)) in Type 1 diabetes mellitus. J Comp Eff Res. 2021 Jun;10(9):763-775. doi: 10.2217/cer-2020-0208. Epub 2021 Apr 30. PMID 33928797